CLINICAL TRIAL: NCT06386198
Title: HEalth Advocate for Liver Transplantation: Improving Transition of Care for Adolescent Liver Transplant Recipients
Acronym: HEAL-Tx:ToC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: American Society of Transplantation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-40699
Record Dates: First submitted 2024-04-23; First posted 2024-04-26 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Liver Transplant; Complications; Pediatric ALL
Keywords: Health Advocate; Patient Navigator
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): This is a single arm pilot intervention.
  Interventions: Behavioral: Health Advocate

INTERVENTIONS:
Behavioral: Health Advocate — The Health Advocate intervention will include helping pediatric liver transplant recipients and their families address unmet household social needs (e.g., food insecurity), improve patient-provider communication, and enhance care coordination.
  Other Names: Patient Navigator

SUMMARY:
The Health Advocate for Liver Transplant (HEAL-Tx) Transition of Care Pilot is a nonrandomized, open-label intervention pilot of a health advocate intervention aimed to assess feasibility and acceptability of integrating a Health Advocate onto the transplant team to help adolescents transition their care to adult transplant teams. Across studies, health advocate roles vary, and can include coordinating medical care treatment, facilitating financial assistance (e.g., taxi vouchers), and connecting patients to community resources, which can improve self-management, mitigate social risks, and lead to better communication between the healthcare system and the family. In this pilot, the investigators will adapt this intervention for adolescent/young adult liver transplant patients and measure acceptability and feasibility according to RE-AIM.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has received a liver transplant >1 year ago
2. Study team has screened patient and discussed with the primary transplant practitioner that patient may benefit from the Health Advocate program.
3. Patient has an unmet social risk (e.g., food insecurity) or MLVI >/= 2.0.
4. Patient will be transferred to adult transplant team in <6 months.
5. Patient can read and write English or Spanish
6. Patient is between 18-25 years old and can provide informed consent.
7. Patient has a working phone and smart device capable of video and/or audio virtual visits via Zoom.

Exclusion Criteria:

* Patient has significant cognitive impairment.
* Does not meet age criteria
* Patient is a ward of the state.
* Non-English, non-Spanish speakers.
* Non-US residents.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-03 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in patient experience | Baseline and 180 days
  The investigators will administer a survey of patient experience at study enrollment and at the end of the intervention to assess for changes in patient experience with the transplant team. These questions will focus on experiences receiving transplant care, experiences discussing social needs with the transplant team, and overall subjective assessment of the transplant recipient's overall health.

SECONDARY OUTCOMES:
Change in medication adherence using MLVI | Baseline and 180 days
  Medication level variability index (MLVI) defined as the standard deviation of at least 3 outpatient tacrolimus trough levels (binary >/=2.0 or <2.0). The investigators will assess this at study entry and again at 180 days.
The quality of health advocate interactions with the participants, healthcare team, and community-based resources. | 180 days
  The Health Advocate will keep a detailed journal entry after each encounter and certain Health Advocate interactions will be recorded. The investigators will qualitatively analyze these journal entries and recordings to identify what functions the health advocate undertook.
A qualitative assessment of patient and healthcare provider satisfaction with the Health Advocate intervention. | 180 days
  The investigators will conduct in-depth interviews with the patient participant and clinical team members to assess overall satisfaction with the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Sharad Wadhwani, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of California San Francisco, San Francisco, California
  - Children's Healthcare of Atlanta, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No